CLINICAL TRIAL: NCT04453904
Title: A Multicenter Randomized Controlled Study of Modalities of Adjuvant Radiotherapy and Chemotherapy for Stage Ⅲ Endometrial Cancer
Brief Title: Modality of Adjuvant Radiotherapy and Chemotherapy for Stage Ⅲ Endometrial Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020PHB013-01
Record Dates: First submitted 2020-03-16; First posted 2020-07-01 (Actual); Last update posted 2020-07-01 (Actual); Status verified 2020-06

CONDITIONS: Endometrial Cancer
Keywords: radiochemotherapy; sanwich mode
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- sequential radiochemotherapy in a "sanwich" mode (Experimental): Two courses of TC regimen chemotherapy (paclitaxel 135-175mg / m2; carboplatin AUC = 5; once every 21 days) will be given first, followed by external pelvic radiation (± vaginal brachytherapy), and then four courses of the same regime consolidation chemotherapy.
  Interventions: Other: sequential radiochemotherapy in a "sanwich" mode
- concurrent chemoradiotherapy followed by chemotherapy (Active Comparator): External pelvic radiation (± vaginal brachytherapy) will be given after operation. On the first day and the 29th day of radiotherapy, concurrent intravenous cisplatin (50mg/m2) will be given. After the concurrent radiochemotherapy, four courses of TC regimen (paclitaxel 135-175mg / m2; carboplatin AUC = 5; once every 21 days) chemotherapy will be given.
  Interventions: Other: sequential radiochemotherapy in a "sanwich" mode

INTERVENTIONS:
Other: sequential radiochemotherapy in a "sanwich" mode — Patients will randomized into two different modalities of radiochemotherapy.

SUMMARY:
Endometrial cancer is the most common gynecological malignancy affecting women's health. About 15% of the patients will have local late disease (stage III) with high risk of recurrence and tumor related mortality. There is a consensus that adjuvant radiochemotherapy is needed for stage Ⅲ endometrial cancer, but the best modality of radiochemotherapy is still uncertain. The retrospective data of our center showed that the sequential radiochemotherapy of "chemotherapy-radiotherapy-chemotherapy" in the "sanwich" mode could improve the survival outcome in patients with advanced endometrial cancer. A multicenter, prospective, randomized controlled study to compare the "sanwich" mode of radiochemotherapy and the "concurrent chemoradiotherapy followed by chemotherapy" mode will be carried out to determine the better modality of radiochemotherapy in stage III endometrial adenocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. patients of primary treatment
2. All patients must have undertaken comprehensive staging operation（Surgery must have included a hysterectomy and bilateral salpingooophorectomy and surgical staging).
3. Patients with endometrial adenocarcinoma confirmed by postoperative patholog.
4. All patients with Surgical Stage III endometrial carcinoma according to FIGO 2009 staging criteria.
5. Entry into the study is limited to no more than 8 weeks from the date of surgery.
6. Patients with adequate organ function, reflected by the following parameters:

   1. WBC ≥ Normal value of the institution;
   2. Absolute neutrophil count (ANC) ≥ Normal value of the institution;
   3. Platelet count ≥ 100,000/mcl;
   4. SGOT, SGPT, and alkaline phosphatase ≤ 1.25 X upper limit of normal (ULN) ;
   5. Bilirubin ≤ 1.5 X ULN;
   6. Creatinine ≤ institutional ULN.
7. Patients with a Karnofsky score≥60.
8. The patients should voluntarily join the study, sign an approved informed consent with good compliance and cooperation with the follow-up.

Exclusion Criteria:

1. Patients who have received prior adjuvant therapy (radiotherapy or chemotherapy or endocrine therapy).
2. Patients with residual tumor after surgery.
3. Patients with other invasive malignancies.
4. Patients with contraindications of radiotherapy and chemotherapy (with a history of myocardial infarction within 3 month, unstable angina pectoris or history of uncontrolled arrhythmia s from the date of registration) and who cannot receive postoperative adjuvant radiotherapy and chemotherapy.
5. Patients with an estimated survival of less than 6 months.
6. Those who are unable or unwilling to comply with the research requirements

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 654 (Estimated)
Dates: Start 2020-05-12 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Progress-free survival | From the date of randomization until the date of first documented progression or date of death from any cause, whichever came first,assessed up to 60 months
  To determine if treatment with radiochemotherapy in "sanwich" mode (carboplatin and paclitaxel for 2 cycles, then radiotherapy, and then carboplatin and paclitaxel for 4 cycles)(experimental arm) reduces the rate of recurrence or death (i.e., increases disease-free survival) when compared to concurrent cisplatin and radiation followed by carboplatin and paclitaxel for 4 cycles (control arm) in patients with stages III endometrial adenocarcinoma.

SECONDARY OUTCOMES:
Overall survival | From the date of randomization until the date of death from any cause, assessed up to 60 months
  To determine if treatment with radiochemotherapy in "sanwich" mode (carboplatin and paclitaxel for 2 cycles, then radiotherapy, and then carboplatin and paclitaxel for 4 cycles)(experimental arm) reduces the rate of death (i.e., increases survival) when compared to concurrent cisplatin and radiation followed by carboplatin and paclitaxel for 4 cycles (control arm) in patients with stages III endometrial adenocarcinoma.
adverse effect | through study completion,an average of 1 year
  To compare the modalities with respect to acute and late adverse effects of therapy.
patient-reported Quality of Life | 3 months after treatment and 1 year after treatment
  To determine the impact on patient-reported Quality of Life (using the questionnaire of combining the items from FACT-G, FACT/GOG-NTX-4 subscale (4 items) and items C3 and C5 from the FACT-C)during and following treatment for up to 1 year with the two treatment regimens.

CONTACTS AND LOCATIONS:
Locations (1):
- Jianliu Wang, Beijing, Beijing Municipality, China